CLINICAL TRIAL: NCT00006387
Title: A Phase I Study of RAS Peptide Vaccination in Patients With Advanced Pancreatic or Colorectal Adenocarcinoma
Brief Title: Vaccine Therapy Plus QS21 in Treating Patients With Advanced Pancreatic or Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: FCCC-98026; NCI-T97-0051 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2000-10-04; First posted 2004-06-09 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer; Pancreatic Cancer
Keywords: stage IV colon cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — saponin QA-21V1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: QS21
Biological: ras peptide cancer vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. QS21 may improve the ability of the immune system to respond to disease. Combining vaccine therapy with QS21 may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy plus QS21 in treating patients who have advanced pancreatic or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of ras peptide cancer vaccine plus immunological adjuvant QS21 in patients with advanced pancreatic or colorectal adenocarcinoma. II. Determine the immunologic effects of this treatment regimen in these patients. III. Determine the antitumor effect of this treatment regimen in these patients.

OUTLINE: This is a dose escalation study of ras peptide cancer vaccine. Patients receive ras peptide cancer vaccine mixed with immunological adjuvant QS21 subcutaneously monthly for 4 doses, every 2 months for 4 doses, every 4 months for 3 doses, every 6 months for 2 doses, and then annually thereafter in the absence of unacceptable toxicity. Cohorts of 3 to 6 patients receive escalating doses of ras peptide cancer vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 4 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 15-20 patients will be accrued for this study within 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced pancreatic or colorectal adenocarcinoma Curatively unresectable OR Recurrent following potentially curable resection OR Pancreatic adenocarcinoma that has been surgically resected within the past 12 months Must have one of the following ras gene mutations at codon 12: Glycine to cysteine Glycine to aspartic acid Glycine to valine HLA A2 required if evidence of HLA restriction for peptide presentation

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,500/mm3 Lymphocyte count at least 500/mm3 Hepatic: Bilirubin no greater than 3 mg/dL Renal: Creatinine no greater than 2 times upper limit of normal OR Creatinine clearance at least 50 mL/min Other: No active infection requiring sytemic therapy No history of severe allergy or anaphylaxis No immunodeficiency (e.g., HIV infection, lupus, or myeloma) Not pregnant Negative pregnancy test Fertile patients must use effective contraception Women must use contraception for 3 months prior to, during and for 3 months after study Men must use contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunologic therapy No other concurrent systemic immunotherapy for cancer Chemotherapy: At least 4 weeks since prior chemotherapy No concurrent systemic chemotherapy for cancer Endocrine therapy: At least 4 weeks since prior corticosteroids No concurrent corticosteroids Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Other: At least 4 weeks since prior immunosuppressants (e.g., methotrexate) No concurrent immunosuppressants Concurrent nonsteroidal antiinflammatory drugs for pain palliation allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2000-10; Primary Completion 2002-01 (Actual); Study Completion 2002-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal J. Meropol, MD, Study Chair — Fox Chase Cancer Center